CLINICAL TRIAL: NCT05127096
Title: Sample Collection Study for the CellMax Life Circulating Tumor Cell and Circulating Tumor DNA Platforms for the Early Detection of Colorectal Cancer and Adenomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CellMax Life (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO00100
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Colorectal Cancer Screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cohort A: Cohort A will include subjects with a recent diagnosis of colorectal cancer and/or advanced adenoma requiring additional endoscopic or surgical resection (surgery).
  Interventions: Diagnostic Test: FirstSight blood test
- Cohort B: Cohort B will include subjects undergoing routine screening colonoscopies will be enrolled in the screening cohort.
  Interventions: Diagnostic Test: FirstSight blood test

INTERVENTIONS:
Diagnostic Test: FirstSight blood test — FirstSight blood test for colorectal cancer screening

SUMMARY:
The purpose of this study is to collect clinical specimens from subjects with a diagnosis of colorectal cancer/advanced adenoma or undergoing a screening colonoscopy and meeting study eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

To enroll in Cohort A, a subject must:

* Be 45-80 years of age (inclusive) at the time of screening.
* Be recently diagnosed with primary colorectal cancer or advanced adenoma with plans to surgically remove the target lesion.

To enroll in Cohort B, a subject must:

* Be 45-80 years of age (inclusive) at the time of screening.
* Be planning to undergo a screening colonoscopy within 30 days after providing signed informed consent.

Exclusion Criteria:

To enroll in Cohort A, a subject must NOT have:

* Inflammatory bowel disease (IBD)
* Personal or family history of colorectal cancer syndromes or other hereditary cancer syndromes

To enroll in Cohort B, a subject must NOT have:

* Personal history of colorectal cancer, colorectal adenoma or aerodigestive tract cancer.
* Personal or family history of Familial adenomatous polyposis (FAP).
* Personal or family history of Hereditary non-polyposis colorectal cancer syndrome (HNPCC or Lynch Syndrome).
* Positive fecal occult blood testing (FOBT) within the previous 6 months.
* Positive fecal immunochemical testing (FIT) in the previous 6 months.
* Colorectal resection for any reason other than sigmoid diverticular disease.
* Overt rectal bleeding within the previous 30 days.
* Personal history of any cancer diagnosed <5 years prior.
* Inflammatory bowel disease (IBD), including chronic ulcerative colitis (CUC) and Crohn's disease.
* Colonoscopy within the previous 9 years.
* Barium enema, computed tomographic colonography, or sigmoidoscopy within the previous 5 years.
* ≥ 2 first-degree relatives who have been diagnosed with colorectal cancer (Note: First degree relatives include parents, siblings and offspring).
* 1 first-degree relative with CRC diagnosed before the age of 60.
* Have participated or be currently participating in a clinical research study in which an experimental medication has been administered during the 30 days up to and including the date of providing informed consent or may be administered through the time of the colonoscopy.
* Have a medical condition which, in the opinion of the investigator, should preclude enrollment into the study.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort A: This cohort will include subjects with a recent diagnosis of colorectal cancer or advanced adenoma requiring surgical resection.
  Cohort B: This cohort will include subjects undergoing routine screening colonoscopies for colorectal cancer as part of their regular medical assessment regimen.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity for CRC of the FirstSight test | 30 days
Specificity of the FirstSight test | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Rui Mei, PhD, Study Director — CellMax Life
Locations (15):
- United States (15):
  - CellMax Site A, Huntsville, Alabama
  - CellMax Site O, Chula Vista, California
  - CellMax Site L, Lancaster, California
  - CellMax Site J, Tustin, California
  - CellMax Site P, Coral Gables, Florida
  - CellMax Site D, Coral Springs, Florida
  - CellMax Site G, Coral Springs, Florida
  - CellMax Site C, Miami, Florida
  - CellMax Site B, Metairie, Louisiana
  - CellMax Site N, Mentor, Ohio
  - CellMax Site M, Camp Hill, Pennsylvania
  - CellMax Site K, Houston, Texas
  - CellMax Site E, McAllen, Texas
  - CellMax Site F, Pasadena, Texas
  - CellMax Site H, San Antonio, Texas